## A Pilot Feasibility and Acceptability Study of a Relational Playbook and Coaching Intervention for Cardiology Teams to Enhance Employee Well-being and Veteran Care

NCT06456021

April 12, 2024



Study Title: Pilot Feasibility and Acceptability Study of a Relational Playbook and Coaching Intervention for Cardiology

Teams to Enhance Employee Well-being and Veteran Care **Primary Investigator:** Name: Heather Gilmartin, PhD, NP

**COMIRB Protocol Number: 17-1153** 

Version date: 04/12/2024

\_\_\_\_\_

You are being asked to be in this research study because you are a Veterans Health Administration (VA) cardiac catheterization laboratory staff member.

If you join this study, you will implement the Relational Playbook for Cardiology Teams and receive either standard implementation support or enhanced implementation support. You will be asked to complete surveys and participate in a recorded interview assessing the intervention.

The study is designed to learn more about the implementation, feasibility, and acceptability of the Relational Playbook, a workforce development intervention, and two implementation support approaches.

Possible discomforts or risks include increased workload during the study and possible loss of confidentiality. There may be risks the researchers have not thought of.

The study is not designed to benefit you directly.

Every effort will be made to protect your privacy and confidentiality. The study team will not disclose participation in the study or responses to any questions to anyone outside the research team. Interviews and coaching sessions will be conducted via VA Teams at a time convenient to the participants, and the notes will be saved directly to an access-controlled data folder on a secure server at VA Eastern Colorado Healthcare System.

This research is being paid for by the VA Office of Research Development – Health Systems Research Pilot Investigator Initiated Award mechanism.

You have a choice about being in this study. You do not have to be in this study unless you want to be.

The data we collect will be used for this study but may also be important for future research. Your data may be used for future research or distributed to other researchers for future study without additional consent if information that identifies you is removed from the data.

If you have any questions, you can call Heather Gilmartin, PhD, NP at xxx-xxx. You can call to ask questions at any time.

You may have questions about your rights as someone in this study. If you have questions, you can call COMIRB (the responsible Institutional Review Board) at 303-724-1055.